CLINICAL TRIAL: NCT02311101
Title: Sequential Intravesical Mitomycin Plus Bacillus Calmette-Guérin for Non-Muscle Invasive Urothelial Bladder Carcinoma: Translational and Phase I Clinical Trial
Brief Title: Phase I Mitomycin Combined With Bacillus Calmette-Guérin (BCG) for Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Robert Svatek, Assistant Professor, Division of Urologic Oncology, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20120003H
Record Dates: First submitted 2013-04-14; First posted 2014-12-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Urinary Bladder Neoplasm
Keywords: bladder cancer; mitomycin; BCG; intravesical; non-muscle invasive
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Therapy Group MMC 10/BCG Half (Experimental): Intravesical Mitomycin C and intravesical BCG
  First intravesical mitomycin C (10 mg) is instilled for 30 minutes. Then the mitomycin is removed and the bladder is gently hand-irrigated with sterile water for 15 minutes in order to facilitate removal of mitomycin C. Then, intravesical BCG (half dose) is instilled for 2 hours under usual conditions. Full dose BCG corresponds to 1 to 8x10^8 colony-forming units of BCG. This study targets patients with BCG-naive or BCG-refractory high-risk non-muscle invasive bladder cancer. The first 3 participants received 10mg of MMC and half dose of BCG. The dose was assigned in order of enrollment.
  Interventions: Drug: Mitomycin C
- Therapy Group MMC 10/BCG Full (Experimental): First intravesical mitomycin C (10 mg) is instilled for 30 minutes. Then the mitomycin is removed and the bladder is gently hand-irrigated with sterile water for 15 minutes in order to facilitate removal of mitomycin C. Then, intravesical BCG (full dose) is instilled for 2 hours under usual conditions. Full dose BCG corresponds to 1 to 8x10^8 colony-forming units of BCG. This study targets patients with BCG-naive or BCG-refractory high-risk non-muscle invasive bladder cancer. The following 3 participants received 10mg of MMC and full dose BCG. Dose was assigned in order of enrollment.
  Interventions: Drug: Mitomycin C
- Therapy Group MMC 20/BCG Full (Experimental): First intravesical mitomycin C (20 mg) is instilled for 30 minutes. Then the mitomycin is removed and the bladder is gently hand-irrigated with sterile water for 15 minutes in order to facilitate removal of mitomycin C. Then, intravesical BCG (full dose) is instilled for 2 hours under usual conditions. Full dose BCG corresponds to 1 to 8x10^8 colony-forming units of BCG. This study targets patients with BCG-naive or BCG-refractory high-risk non-muscle invasive bladder cancer. The next 3 participants enrolled received 20mg of MMC and full dose BCG. Dose was assigned in order of enrollment.
  Interventions: Drug: Mitomycin C
- Therapy Group MMC 40/BCG Full (Experimental): First intravesical mitomycin C (40 mg) is instilled for 30 minutes. Then the mitomycin is removed and the bladder is gently hand-irrigated with sterile water for 15 minutes in order to facilitate removal of mitomycin C. Then, intravesical BCG (full dose) is instilled for 2 hours under usual conditions. Full dose BCG corresponds to 1 to 8x10^8 colony-forming units of BCG. This study targets patients with BCG-naive or BCG-refractory high-risk non-muscle invasive bladder cancer. The last 3 participants received 40mg of MMC and full dose BCG. Dose was assigned in order of enrollment.
  Interventions: Drug: Mitomycin C

INTERVENTIONS:
Drug: Mitomycin C — Given intravesically
  Other Names: BCG

SUMMARY:
The study aims to establish the safety and toxicity of a combined intravesical mitomycin C with BCG for patients with bladder cancer.

DETAILED DESCRIPTION:
Urine Sample Collection and Handling: Voided urine will be collected pre and post BCG procedure. Urinalysis will be performed if participant presents with urinary symptoms. Analysis of urinary cytokines as predictors of response to therapy will be conducted by ELISA kits.

Tissue Sample Collection and Handling: Tissue biopsy specimens will be collected pre BCG procedure. Analysis of gene expression will be conducted.

TEST PROCEDURES Subjects will be given one of three concentrations of Mitomycin C (MMC) (10 mg in 20 mL, 20 mg in 20 ml or 40 mg in 20 ml) for 30 minutes followed by a 10 minute washout period. Followed by three concentrations of BCG including ¼ strength, ½ strength, and full strength for 2 hours. Dose escalation will take place among subsequent patients and not within each patient.

Approximately 30 subjects will be enrolled to reach the target completion enrollment of 10 subjects.

Long-term Follow-up A Chart review will be conducted every three months for 2 years after initial 6 month study data collection. Patient charts will be reviewed to assess disease progression and any data supporting findings. Long-term follow-up is necessary to determine recurrence rates and long-term safety and efficacy of Mitomycin/BCG treatment therapy as well as BCG therapy in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or recurrent multi-focal Ta, large Ta, high-grade Ta, CIS, or T1 bladder cancer
2. In urologist's opinion a good candidate for BCG induction therapy
3. Be able to give informed consent
4. Be age 18 or older.

Exclusion Criteria:

1. Inadequate marrow function (defined as granulocytes less than 1,500 cells/mm3 and platelets less than 150,000 cells/mm3)
2. Immunosuppressed state (e.g. HIV, use of chronic steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 3 months
  The primary objective of this study is to determine the MTD for sequential MMC with BCG and thereby establish a recommended phase 2 dose of the combined therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Svatek, MD, MSCI, Principal Investigator — UT Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Hilton WM, Ercole B, Parekh DJ, Sonpavde G, Ghosh R, Svatek RS. Efficacy of combined intravesical immunotherapy and chemotherapy for non-muscle invasive bladder cancer. Expert Rev Anticancer Ther. 2011 Jun;11(6):949-57. doi: 10.1586/era.11.69. PMID 21707292